CLINICAL TRIAL: NCT00997698
Title: Imaging Epidemiological Investigation of Intracranial Aneurysms and the Prospective Study of Risk Factors：Assessment of MR Imaging Trail
Brief Title: Contrast-enhanced Magnetic Resonance Angiography Investigation of Intracranial Aneurysms and Prospective Study of Risk Factors
Acronym: EIIA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Military Medical University (Other)
Responsible Party: Changhai Hospital affiliated to Second Military Medical University, Changhai Hospital affiliated to Second Military Medical University
Other Study IDs: SecondMMU
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm; Magnetic resonance angiography; Epidemiology
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective observational registry with intent to detect the prevalence of intracranial aneurysms with contrast-enhanced MR angiography (CE-MRA) at 1.5T, and to determine the risk factors such as high blood pressure and cigarette smoking relating to intracranial aneurysms.

DETAILED DESCRIPTION:
Intracranial aneurysms are common and have been reported increased incidence rate because of the widespread use of high-resolution imaging techniques. They are clinically important because of the life-threatening rupture and hemorrhage. Early detection and diagnosis is the key of treatment. Contrast-enhanced MR angiography (CE-MRA), as a simple, sensitivity and noninvasive method, is playing an important role in Vascular Imaging. CE-MRA has been an accuracy modality for intracranial aneurysm at most centers and proved the high sensitivity and accuracy comparing with DSA. Therefore, we use CE-MRA at 1.5T as a tool of epidemiological investigation of intracranial aneurysms.

In retrospective analysis, conventional risk factors for intracranial aneurysms include hypertension, hyperlipidemia, diabetes mellitus (DM), smoking history, and family history, etc. However, retrospective analysis probably gives an underestimation or overestimation of the actual results. Prospective analysis will get accurate data on the risk factors relating to intracranial aneurysms

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 80 years
* Willing to undergo study procedures
* Who are fully informed about the study and have signed the informed consent form

Exclusion Criteria:

* History of intracranial aneurysm
* History of intracranial tumor
* History of cerebral infarction
* Acute stroke
* Require emergency treatment
* Contraindication for MRI examination
* Severely impaired renal functions
* Known anaphylactic reaction to MR contrast media
* Pregnancy or nursing

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People coming to Changhai hospital to get health check or consult docter, undergoing cerebral CE-MRA, and according with the criteria were recruited. Assuming an 8 percent prevalence of intracranial aneurysm in the general population and using a two-sided alpha value of 0.05, we estimated that 4000 persons would need to be enrolled for the study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Intracranial aneurysms identified by CE-MRA | 24 months

SECONDARY OUTCOMES:
Statistical analysis of the prospective factors which contribute to the development of intracranial aneurysms | 6 months after the study

CONTACTS AND LOCATIONS:
Overall Officials: Ping J Lu, MD, PhD, Study Director — Changhai Hospital affiliated to Second Military Medical University; Qi Liu, MD, PhD, Principal Investigator — Changhai Hospital affiliated to Second Military Medical University
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China